CLINICAL TRIAL: NCT07096011
Title: Studying Phenotypic Risks for Obesity and Underlying Traits in Young Infants: A Pilot Study
Brief Title: Studying Phenotypic Risks for Obesity and Underlying Traits in Young Infants
Acronym: SPROUT
Status: Recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Emily W. Flanagan, MS, PhD, Principal Investigator, Pennington Biomedical Research Center
Other Study IDs: 2025-026
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Infant Body Composition and Metabolism; Metabolism; Energy Expenditure; Infant Formula; Human Milk, Breast Milk; Metabolic Flexibility
Keywords: infant; metabolism; energy expenditure; infant formula; breast milk; human milk; thrifty phenotype; metabolic flexibility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — human milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Meal Test - Human Milk — Infants will be fed a mixed meal test (meal challenge test) of human milk from his/her human milk donor (e.g., mother). Since all infants enrolled in the study consume human milk as a primary food source, this meal challenge test represents their standard meal, at a larger size. The meal test is provided inside a metabolic chamber to measure energy expenditure (VCO2 and VO2) before and after the meal. The amount of human milk that the infant is fed is estimated using the age and sex specific equations from the 2023 DRI for infants aged 0-2 years. Infants will be provided 20% of their predicted energy needs, which is equivalent to between 4-6 ounces of food for most infants of this age. The caloric content for human milk is be estimated at 20 kcals/ounce.
Other: Meal Test - Infant Formula — Infants will be fed a mixed meal test (meal challenge test) of ready-to-feed infant formula. Since all infants enrolled in the study consume human milk as a primary food source, this meal challenge test represents a meal different from their habitual food intake and is a standard meal that all participants receive. The meal test is provided inside a metabolic chamber to measure energy expenditure (VCO2 and VO2) before and after the meal. The amount of infant formula that the infant is fed is estimated using the age and sex specific equations from the 2023 DRI for infants aged 0-2 years. Infants will be provided 20% of their predicted energy needs, which is equivalent to between 4-6 ounces of food for most infants of this age. The caloric content for the ready-to-feed infant formula is 20 kcals/ounce.

SUMMARY:
The purpose of this research study is to understand how infants metabolize different meals and to develop clinical tools which identify infants as having two different phenotypes. The phenotypes are the 1) metabolic "thriftiness" and 2) the metabolic flexibility.

DETAILED DESCRIPTION:
The purpose of this research study is to understand how infants metabolize different meals and to develop clinical tools which identify infants as having two different phenotypes. This will be accomplished by providing two meal test stimuli to infant participants (human milk and infant formula). Energy expenditure and respiratory exchange ratio will be obtained before and after the meals to calculate the delta in both. From there, two phenotypes will be identified. The first phenotypes is metabolic "thriftiness", which will be defined by the energy expenditure after consuming two standard meals. The second phenotype is the degree of metabolic flexibility and will be defined by substrate oxidation (using respiratory exchange ratio) following two standard meals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 weeks to less than 17 weeks at screening
* Being fed human milk as a primary source of food
* Be willing to consume one meal of infant formula
* Be willing to complete a DXA measurement

Exclusion Criteria:

* Unable to complete the screening visit and two clinic visits within 14 days
* Born with health conditions that would render procedures unsafe
* Born earlier than 35 days and 0 weeks gestation
* Eating supplemental foods
* Physician diagnosed feeding difficulties that may require a special type of nipple for bottle feeding

Ages: 2 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Up to 40 infants who are less than 17 weeks will be recruited to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure difference from baseline to postprandial | 60 minutes
  Percent difference from baseline to postprandial energy expenditure
Energy expenditure difference from baseline to postprandial (2) | 60 minutes
  Absolute difference between baseline and postprandial energy expenditure

SECONDARY OUTCOMES:
Thrifty and Spendthrift Phenotypes | 60 minutes
  Number of infants with a thrifty and spendthrift phenotype
Metabolic flexibility | 60 minutes
  Difference in respiratory exchange ratio from baseline to postprandial

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided